CLINICAL TRIAL: NCT00331630
Title: Pilot Neoadjuvant Trial in Breast Cancer With Combination of ABI-007 (Abraxane) and GW572016 (Lapatinib)
Brief Title: Abraxane and Lapatinib in Treating Patients With Stage I, Stage II, or Stage III Breast Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: GlaxoSmithKline (Industry); Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 05B2; NU 05B2 (Other: Northwestern University); STU00007257 (Other: Northwestern University IRB)
Record Dates: First submitted 2006-05-30; First posted 2006-05-31 (Estimated); Results first posted 2020-03-06 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-01

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Lapatinib; Taxes; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment arm (Experimental): 30 patients receive Abraxane IV over 30 minutes on day 1 and oral lapatinib once daily on days 1-21. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: lapatinib ditosylate; Drug: paclitaxel albumin-stabilized nanoparticle formulation

INTERVENTIONS:
Drug: lapatinib ditosylate — Oral lapatinib is taken once daily on days 1-21 of each treatment cycle. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.
  Other Names: Tykerb; Tyverb
Drug: paclitaxel albumin-stabilized nanoparticle formulation — 30 patients receive Abraxane IV over 30 minutes on day 1 each of each treatment cycle. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.
  Other Names: Abraxane; ABI-007

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as Abraxane, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Lapatinib may stop the growth of tumor cells by blocking some of the enzymes needed for their growth. Giving Abraxane together with lapatinib may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving Abraxane together with lapatinib works in treating patients with stage I, stage II, or stage III breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the clinical response rate, as measured by clinical exam and imaging studies, in patients with stage I-III breast cancer treated with neoadjuvant Abraxane in combination with lapatinib.

Secondary

* Determine the pathologic complete response rate in patients treated with this regimen.
* Correlate proliferation (Ki67), apoptosis (cleaved caspase-3), and angiogenesis (vW, CD34) markers, measured before and after treatment, with tumor response in these patients.
* Conduct other correlative studies, including epidermal growth factor receptor (EGFR), HER2/neu, matrix metalloproteinases (MMPs), and transforming growth factor (TGF-β), before and after treatment with this regimen to assess tumor response in these patients.
* Determine the toxicity of this regimen in these patients.

OUTLINE: This is a pilot study. Patients are assigned to 1 of 2 treatment groups.

* Group 1: The first 10 patients receive Abraxane IV over 30 minutes on day 1 and oral lapatinib once daily on days 1-21. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.
* Group 2: The next 20 patients receive Abraxane and lapatinib (at a higher dose) as in group 1. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.

Patients undergo blood collection and tumor biopsies periodically for correlative biomarker studies.

PROJECTED ACCRUAL: A total of 30 patients will be accrued to this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed breast cancer

  * Clinical stage I-III disease
* Measurable disease defined as ≥ 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques OR ≥ 10 mm with spiral CT scan
* HER2/neu 3+ by immunohistochemistry or positive by fluorescent in situ hybridization
* No known brain metastases
* Hormone receptor status unspecified

PATIENT CHARACTERISTICS:

* Menopausal status not specified
* Male or female
* Life expectancy > 12 weeks
* ECOG performance status (PS) 0-1 OR Karnofsky PS 80-100%
* WBC ≥ 3,000/mm^3
* Absolute neutrophil count ≥ 1,500 mm^3
* Platelet count ≥ 100,000/mm^3
* Total bilirubin normal
* AST and ALT ≤ 2.5 times upper limit of normal
* Creatinine normal OR creatinine clearance ≥ 60 mL/min
* LVEF ≥ 50% as measured by echocardiogram or MUGA scan
* No other malignancy within the past year
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Able to swallow and retain oral medication
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to lapatinib
* No ongoing or active infection
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* No psychiatric illness or social situation that would preclude study compliance
* No other uncontrolled illness
* No gastrointestinal (GI) tract disease that would preclude ability to take oral medication
* No malabsorption syndrome
* No requirement for IV alimentation
* No uncontrolled inflammatory GI disease (e.g., Crohn's disease or ulcerative colitis)

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy, immunotherapy, radiotherapy, or hormonal therapy for breast cancer
* No prior treatment with epidermal growth factor receptor targeting therapies
* No prior surgical procedures affecting absorption
* No prior surgery for breast cancer
* At least 14 days since prior and no concurrent CYP3A4 inducers, including any of the following:

  * Dexamethasone or dexamethasone equivalent dose ≥ 1.5 mg/day, including any of the following:

    * Cortisone (≥ 50 mg/day)
    * Hydrocortisone (≥ 40 mg/day)
    * Prednisone (≥ 10 mg/day)
    * Methylprednisolone (≥ 8 mg/day)
  * Phenytoin
  * Carbamazepine
  * Phenobarbital
  * Efavirenz
  * Nevirapine
  * Rifampin
  * Rifabutin
  * Rifapentine
  * Hypericum perforatum (St. John's wort)
  * Modafinil
* At least 7 days since prior and no concurrent CYP3A4 inhibitors, including any of the following:

  * Clarithromycin
  * Erythromycin
  * Troleandomycin
  * Delavirdine
  * Ritonavir
  * Indinavir
  * Saquinavir
  * Nelfinavir
  * Amprenavir
  * Lopinavir
  * Itraconazole
  * Ketoconazole
  * Voriconazole
  * Fluconazole (doses up to 150 mg/day are permitted)
  * Nefazodone
  * Fluvoxamine
  * Verapamil
  * Diltiazem
  * Cimetidine
  * Aprepitant
  * Grapefruit or its juice
* At least 6 months since prior and no concurrent amiodarone
* At least 2 days since prior and no concurrent gastric pH modifiers*, including any of the following:

  * Cimetidine
  * Ranitidine
  * Nizatidine
  * Famotidine
  * Omeprazole
  * Esomeprazole
  * Rabeprazole
  * Pantoprazole
  * Lansoprazole
* NOTE: *Antacids are allowed within 1 hour before and after administration of study drug
* No other concurrent investigational agents
* No other concurrent anticancer therapy, including chemotherapy, radiotherapy, immunotherapy, or antitumor hormonal therapy
* No concurrent herbal (alternative) medicines
* No concurrent combination antiretroviral therapy for HIV-positive patients
* Concurrent bisphosphonates allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-05-04 (Actual); Primary Completion 2006-11-10 (Actual); Study Completion 2010-08-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Virginia G. Kaklamani, MD, Principal Investigator — Northwestern University
Locations (5):
- United States (5):
  - Northwestern University, Northwestern Medical Faculty Foundation, Chicago, Illinois
  - Hematology-Oncology Associates of Illinois, Chicago, Illinois
  - Midwest Center for Hematology/Oncology, Joliet, Illinois
  - Saint James Hospital and Health Centers Comprehensive Cancer Institute - Olympia Fields, Olympia Fields, Illinois
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas

REFERENCES:
- [Result] Kaklamani VG, Siziopikou K, Scholtens D, Lacouture M, Gordon J, Uthe R, Meservey C, Hansen N, Khan SA, Jeruss JS, Bethke K, Cianfrocca M, Rosen S, Von Roenn J, Wayne J, Parimi V, Jovanovic B, Gradishar W. Pilot neoadjuvant trial in HER2 positive breast cancer with combination of nab-paclitaxel and lapatinib. Breast Cancer Res Treat. 2012 Apr;132(3):833-42. doi: 10.1007/s10549-011-1411-8. Epub 2011 Feb 27. PMID 21359953

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was opened to accrual May 4th 2006 with the first patient being treated on November 10th 2006. 30 patients were enrolled and treated on the study with the study being closed to new enrollment on June 10th 2009 having reached its accrual goal.
Period: Treatment on Study
Arm/Group | Treatment Arm
Started | 30
Completed 1st Cycle | 30
Completed 4 Cycles | 30
Completed | 30
Not Completed | 0
Period: Evaluated for and Completed SOC Surgery
Arm/Group | Treatment Arm
Started | 30
Completed | 28
Not Completed | 2
Not completed — Progressive Disease | 1
Not completed — Lost to Follow-up | 1
Period: Follow up for 5 Years
Arm/Group | Treatment Arm
Started (All patients that are treated on the study go into follow up period.) | 29 (One patient did not enter follow up as was lost to follow up)
Completed | 0
Not Completed | 29
Not completed — Death | 5
Not completed — Data collection was stopped | 24

BASELINE CHARACTERISTICS:
Groups:
- Treatment With Lapatinib and Abraxane: 30 patients receive Abraxane IV over 30 minutes on day 1 and oral lapatinib once daily on days 1-21. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.
  lapatinib ditosylate: Oral lapatinib is taken once daily on days 1-21 of each treatment cycle. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.
  paclitaxel albumin-stabilized nanoparticle formulation: 30 patients receive Abraxane IV over 30 minutes on day 1 each of each treatment cycle. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.
Arm/Group | Treatment With Lapatinib and Abraxane
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response Rate (cRR)
Description: cRR measured by RECIST for target lesions assessed by clinical exam+ mammogram+ ultrasound (US). cRR is defined as number of patients who's best response in any of the assessments (clinical exam/mammogram/US) is CR+PR. Response will be defined as one of the following in either clinical exam, mammogram or US: Complete Response (CR)-Disappearance of all target lesions. Partial Response (PR)>=30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum.
  Stable Disease-neither sufficient shrinkage to qualify for Partial disease nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum LD while on study.
  Progressive Disease <=20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: At Baseline, then before each treatment cycle begins and after 4 cycles of study treatment (1 cycle = 21 days)
Population: One patient did not have an ultrasound after 4 cycles of treatment prior to surgery
Measure: Number; unit: participants
Arm/Group | Treatment With Lapatinib and Abraxane
Number analyzed (Participants) | 29
participants
  Complete Response | 6
  Partial Response | 18
  Stable Disease | 5
  Progressive Disease | 0
  Clinical Response Rate | 24

2. Secondary Outcome: Pathologic Complete Response (pCR)
Description: Pathologic Complete Response (pCR) will be assessed by breast biopsy at baseline and after 4 cycles of study treatment (1 cycle = 21 days) and at surgery. This will be defined as the number of patients that show a pCR after surgery. pCR is defined as the absence of histologic evidence of invasive tumor cells in the surgical breast specimen and axillary lymph nodes.
Time Frame: At baseline, then after 4 cycles of study treatment (1 cycle = 21 days ) and at surgery
Population: One patient did not have an ultrasound after 4 cycles of treatment prior to surgery and one patient was lost to follow up before undergoing surgery
Measure: Number; unit: Count of Participants
Arm/Group | Treatment With Lapatinib and Abraxane
Number analyzed (Participants) | 28
Count of Participants | 5

3. Secondary Outcome: Proliferation (Ki67) Measured at Baseline and After Completion of Study Treatment
Description: Correlation of proliferation (Ki67) will be assessed by breast biopsy at baseline and after 4 cycles of study treatment (1 cycle = 21 days). Ki67 scoring was performed based on degree of staining (0= no staining, 1=weak nuclear staining, 2=moderate nuclear staining, 3=strong nuclear staining). Ki67 scores were counted on a maximum of 10 randomly selected x40 high-power fields with an eyepiece grid of 10x10 squares containing representative sections of tumor and calculated as percentage of positively stained cells to total tumor cells (Percent Score method) Ki67 labeling Index (LI) as assessed by counting a maximum of 1,000 malignant cells at x400 magnification.
Time Frame: At baseline, then after 4 cycles of study treatment (1 cycle = 21 days )
Measure: Mean (Standard Deviation); unit: Labeling Index
Arm/Group | Treatment With Lapatinib and Abraxane
Number analyzed (Participants) | 30
Labeling Index
  Ki67 pre-treatment | 31.56 (14.47)
  Ki67 post-treatment | 30.66 (19.86)
  Ki67 Difference | -1.84 (21.8)

4. Secondary Outcome: Apoptosis (Cleaved Caspase-3) Measured at Baseline and After Completion of Study Treatment
Description: Apoptosis/cleaved caspase-3 (CC3) will be assessed by breast biopsy at baseline and after 4 cycles of study treatment (1 cycle = 21 days). Scoring was based on the degree of staining (0=more than 90% of tumor cells with no staining, 1= more than 90% of tumor cells have weak staining, 2= more than 90% of tumor cells have moderate staining, 3= more than 90% of tumor cells have strong staining). CC3 scores were counted on a maximum of 10 randomly selected x40 high-power fields with an eyepiece grid of 10x10 squares containing representative sections of tumor and calculated as percentage of positively stained cells to total tumor cells (Percent Score method) CC3 labeling Index (LI) as assessed by counting a maximum of 1,000 malignant cells at x400 magnification.
Time Frame: At baseline, then after 4 cycles of study treatment (1 cycle = 21 days )
Measure: Mean (Standard Deviation); unit: Labeling Index
Arm/Group | Treatment With Lapatinib and Abraxane
Number analyzed (Participants) | 30
Labeling Index
  CC3 Pre-treatment | 84.32 (28.21)
  CC3 Post-treatment | 76.58 (29.51)
  CC3 Difference | -5.26 (35.81)

5. Secondary Outcome: Angiogenesis (vW, CD34) Markers as Measured at Baseline and After Completion of Study Treatment
Description: Angiogenesis (vW, CD34) markers will be assessed by breast biopsy at baseline and after 4 cycles of study treatment (1 cycle = 21 days). Expressions were analyzed by light microscopy in invasive breast cancer regions.
  Tumor cells were assigned a score:
  0 = no staining
  1. weak staining less than 1% of tumor cells
  2. = medium staining in 1-10% of tumor cells/weak staining in less than 1% of tumor cells
  3. = medium or strong staining in more than 10% of the tumor cells. Capillary density was assessed in breast sections stained for CD34 at a x200 magnification by counting the number of capillaries per field with five fields per slide and results expressed as the average number of capillaries per field.
Time Frame: At baseline, then after 4 cycles of study treatment (1 cycle = 21 days )
Measure: Mean (Standard Deviation); unit: average number of capillaries per field
Arm/Group | Treatment With Lapatinib and Abraxane
Number analyzed (Participants) | 30
average number of capillaries per field
  CD34 Pre-treatment | 59.54 (17.56)
  CD34 Post-treatment | 73.12 (32.83)
  CD34 Difference | 14.69 (33.47)
  vWF Pre-treatment | 43.11 (22.33)
  vWF Post-treatment | 49.45 (25.33)
  vWF Difference | 4.79 (26.07)

6. Secondary Outcome: Epidermal Growth Factor Receptor (EGFR), and Matrix Metalloproteinases (MMPs), Measured at Baseline and After Completion of Study Treatment
Description: Epidermal growth factor receptor (EGFR), HER2/neu, matrix metalloproteinases (MMPs), and transforming growth factor (TGF-β) will be assessed by breast biopsy at baseline and after 4 cycles of study treatment (1 cycle = 21 days) with expressions analyzed by light microscopy in invasive breast cancer regions.
  MMP2 cytoplasmic staining intensity was assigned a score:
  0=no reactivity,
  1. =1-10% of tumor cells reactive,
  2. =11-25% of tumor cells reactive,
  3. = 26-50% of cells reactive,
  4. = more than 50% of cells reactive
  Greater than or equal to 2+ score was considered positive for expression.
  EGFR membrane staining was assigned a score:
  0 = no staining or faint staining in less than 10% of cells
  1. = faint incomplete membrane staining in more than 10% of cells
  2. = weak to moderate complete membrane staining of more than 10% of cells
  3. = strong complete membrane staining in more than 10% of tumor cells
Time Frame: At baseline, then after 4 cycles of study treatment (1 cycle = 21 days )
Population: Data for HER2/neu and transforming growth factor (TGF-β) was not collected or analyzed.
Measure: Number; unit: participants
Arm/Group | Treatment With Lapatinib and Abraxane
Number analyzed (Participants) | 30
participants
  EGFR 0 : Pre-treatment | 21
  EGFR 0 : Post-treatment | 18
  EGFR 1+ : Pre-treatment | 5
  EGFR 1+ : Post-treatment | 3
  EGFR 2+ : Pre-treatment | 0
  EGFR 2+ : Post-treatment | 0
  EGFR 3+ : Pre-treatment | 0
  EGFR 3+ : Post-treatment | 0
  EGFR 4+ : Pre-treatment | 0
  EGFR 4+ : Post-treatment | 0
  MMP-2 0 : Pre-treatment | 3
  MMP-2 0 : Post-treatment | 2
  MMP-2 1+ : Pre-treatment | 13
  MMP-2 1+ : Post-treatment | 10
  MMP-2 2+ : Pre-treatment | 3
  MMP-2 2+ : Post-treatment | 2
  MMP-2 3+ : Pre-treatment | 1
  MMP-2 3+ : Post-treatment | 1
  MMP-2 4+ : Pre-treatment | 8
  MMP-2 4+ : Post-treatment | 4

7. Secondary Outcome: Side Effects From the Combination of Abraxane and Lapatinib
Description: Side effects from the combination of Abraxane and Lapatinib will be assessed using CTCAE 3.0. Side effects that were related to study treatment and grade 3 or higher were collected where:
  Grade 1= Mild Grade 2 = Moderate Grade 3 = Severe Grade 4 = Life-threatening Grade 5 = Death
Time Frame: At baseline, then before the start of each study treatment cycle (1 cycle = 21 days) begins
Measure: Number; unit: participants
Arm/Group | Treatment With Lapatinib and Abraxane
Number analyzed (Participants) | 30
participants
  Fatigue grade 3 | 2
  Rash | 1
  Diarrhea | 5
  Bone pain | 1
  Pruritus | 1
  Nausea | 1

8. Other Pre Specified Outcome: Circulating Tumor Cell Measurement
Description: Circulating tumor cell measurement will be assessed by lab tests done at baseline, then before each study treatment cycle begins (1 cycle = 21 days)
Time Frame: At baseline, then before each study treatment cycle begins (1 cycle = 21 days)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Patients were followed for 4 cycles of treatment where 1 cycle equals 21 days
Description: Only adverse events that were at least possibly related to the study were recorded and reported on
Arm/Group | Treatment With Lapatinib and Abraxane
All-Cause Mortality (participants affected / at risk) | 5/30
Serious Adverse Events (participants affected / at risk) | 2/30
Other Adverse Events (participants affected / at risk) | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment With Lapatinib and Abraxane (N=30)
Dry Eyes (Eye disorders) | 1 — Also with blurred vision at the time of this event.
Diarrhea (Gastrointestinal disorders) | 1 — Patient also with fatigue, dehydration and pain at the time of the event
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment With Lapatinib and Abraxane (N=30)
Anemia (Blood and lymphatic system disorders) | 8
Leukopenia (Blood and lymphatic system disorders) | 1
Fatigue (General disorders) | 23
Fever (General disorders) | 2
Weight Loss (General disorders) | 2
DERMATOLOGY/SKIN: Dry skin (Skin and subcutaneous tissue disorders) | 4
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 13
Scalp Folliculitis (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 6
Skin Itching (Skin and subcutaneous tissue disorders) | 1
Skin peeling (Skin and subcutaneous tissue disorders) | 1
Rash acne (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 20
GASTROINTESTINAL DISORDERS: Anorexia (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 4
Dehydration (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 22
Dry mouth (Gastrointestinal disorders) | 1
Heartburn/dyspepsia (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 9
Taste alteration(dysgeusia) (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Mucositis/stomatitis (Gastrointestinal disorders) | 3
Infection (Infections and infestations) | 4
Edema (Blood and lymphatic system disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 5
Alkaline Phoshatase Increased (Metabolism and nutrition disorders) | 1
AST/ALT Increased (Metabolism and nutrition disorders) | 1
Bilirubin Increased (Metabolism and nutrition disorders) | 2
Albumin Decreased (Metabolism and nutrition disorders) | 1
Neuropathy:sensory (Nervous system disorders) | 15
Mood alteration - Depression (Psychiatric disorders) | 1
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 2
Head/headache (Nervous system disorders) | 5
Insomnia (Nervous system disorders) | 1
Muscle Pain (Musculoskeletal and connective tissue disorders) | 2
Pain (General disorders) | 2
Bone Pain (General disorders) | 20
Blurred Vision (Eye disorders) | 3
Dry Eyes (Eye disorders) | 2
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No